CLINICAL TRIAL: NCT01999192
Title: A 24-week Phase IIb, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Investigate the Efficacy and Safety of Tregalizumab (BT061) in Combination With Methotrexate in the Treatment of Subjects With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Methotrexate Alone, Followed by a 24-week Extension Phase: T Cell REgulating Arthritis Trial 2b (TREAT 2b)
Brief Title: Study to Investigate the Safety and Efficacy of Tregalizumab in Subjects (MTX-IR) With Active Rheumatoid Arthritis
Acronym: 986
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Biotest (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 986_TREAT 2b; 2013-000114-38 (EudraCT Number); BT986 (Other: Biotest AG)
Record Dates: First submitted 2013-11-17; First posted 2013-12-03 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
Keywords: inadequate response to MTX; Methotrexate; rheumatoid Arthritis; Phase 2b
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tregalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Level 1 Tregalizumab (Experimental): 25mg Tregalizumab s.c. weekly
  Interventions: Drug: Tregalizumab
- Dose Level 2 Tregalizumab (Experimental): 100mg Tregalizumab s.c. weekly
  Interventions: Drug: Tregalizumab
- Dose Level 3 Tregalizumab (Experimental): 200mg Tregalizumab s.c. weekly
  Interventions: Drug: Tregalizumab
- Placebo (Placebo Comparator): Placebo s.c. weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tregalizumab — humanized anti-CD4 mAb
  Other Names: BT061
  Arms: Dose Level 1 Tregalizumab; Dose Level 2 Tregalizumab; Dose Level 3 Tregalizumab
Drug: Placebo — identical end formulation buffer
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of three different Tregalizumab doses in combination with Methotrexate (MTX) in subjects who have active rheumatoid arthritis and an inadequate response to MTX alone.

The overall study duration is 24 weeks followed by a 24 week extension phase.

DETAILED DESCRIPTION:
The planned clinical study 986 (TREAT 2b) is a 24-week study in patients with Active rheumatoid arthritis (RA) who have had an inadequate response to Methotrexate (MTX) alone. The main phase of this study is followed by a 24-week extension phase for subjects meeting the respective entry criteria. Patients will be randomized to one of three different Active treatment groups or Placebo. The primary efficacy variable is the proportion of subjects with an ACR20 response after 12 weeks of double blinded treatment with the study medication based on observed cases in the FAS.

At Week 12, all subjects who had a minimum improvement of at least 20% (from baseline) in their tender joint count (TJC) and swollen joint count (SJC) continued on the same treatment. Subjects who had not demonstrated an improvement of at least 20% of TJC and SJC were assessed as non-responders. Non-responders who received placebo were randomized to an active treatment dose in a blinded manner. Non-responders who received active treatment were rolled up to the next highest dose in a blinded manner, apart from those already on the highest dose. These subjects remained on the highest dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subject demonstrates active RA according to the 1987 American College of Rheumatology (ACR) or 2010 ACR/European League Against Rheumatism (EULAR) classification criteria for RA with functional class I-III for ≥6 months.
2. Subject receives oral or parenteral MTX treatment for ≥12 weeks (overall), with an unchanged mode of application and stable MTX dose of ≥15 mg per week (or ≥12.5 mg per week in case of MTX intolerance), but no more than the highest locally approved dose for RA, for ≥8 weeks prior to baseline. The dose of MTX is expected to remain stable throughout the study and may be adjusted only for safety reasons. If applicable, the dose of folic acid must be unchanged for ≥8 weeks prior to baseline.
3. Subject meets the following two criteria at both screening and baseline: - At least 6 swollen joints at 28-joint assessment. - At least 6 tender joints at 28-joint assessment.
4. Subject has an erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP) above the upper limit of normal (ULN) at screening. These tests may be repeated once during the screening period at the discretion of the investigator.
5. Subject is ≥18 and ≤75 years of age.
6. Subject has a body mass index ≥18 and ≤35 kg/m².
7. Subject receives treatment with corticosteroids ≤10 mg prednisone equivalent, stable for at least 4 weeks prior to baseline and during the study, if applicable.
8. Subject receives treatment with non-steroidal anti-inflammatory drugs (NSAIDs), stable for at least 2 weeks prior to baseline and during the study, if applicable.
9. Female subjects of childbearing potential: has both a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline.
10. Subject is judged to be in good general health as determined by the investigator based upon the results of medical history, laboratory profile, physical examination, chest X-ray (within 3 months before screening date is acceptable), and 12-lead electrocardiogram (ECG).
11. Subject has a cluster of differentiation 4 (CD4) cell count of > 400/µl at screening.

Exclusion Criteria:

1. Subject has previous exposure to any systemic biologic therapy (e.g., etanercept, adalimumab, rituximab, abatacept, tocilizumab), to Janus kinase (JAK) or spleen tyrosine kinase (SYK) inhibitors, or to Tregalizumab. Previous treatment with an anti-TNF agent is allowed only, if all of the following criteria apply: - treatment was stopped for reasons other than lack of efficacy or adverse events (AEs) - treatment was stopped at least 12 weeks or five half-lives of the compound prior to baseline (whichever is longer), and - the treatment period did not exceed 6 weeks.
2. Subject received treatment with conventional disease-modifying anti-rheumatic drugs (DMARDs) apart from MTX in the 12 weeks prior to baseline, and for DMARD leflunomide in the 24 weeks prior to baseline (except where specific leflunomide wash-out procedures were completed, following applicable guidelines).
3. Subject has been treated with intra-articular or parenteral administration of corticosteroids in the 4 weeks prior to baseline. Inhaled corticosteroids for stable medical conditions are allowed.
4. Subject has undergone joint surgery in the 12 weeks prior to baseline (at joints to be assessed within the study) or has undergone major surgery (e.g., abdominal surgery) in the 8 weeks prior to baseline.
5. Subject has a history of acute inflammatory joint disease of an origin other than RA or subject has any other rheumatic disease other than RA (e.g., mixed connective tissue disease, seronegative spondylarthropathy, psoriatic arthritis, Reiter's syndrome, fibromyalgia, systemic lupus erythematosus or any arthritis with onset prior to age 17 years). However, subjects may have secondary Sjögren's syndrome.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald van Vollenhoven, Prof. MD, Principal Investigator — Karolinska Universitetssjukhuset, Solna
Locations (84):
- United States (8):
  - Study Site 07, Paradise Valley, Arizona
  - Study Site 01, Springfield, Illinois
  - Study Site 03, Lincoln, Nebraska
  - Study Site 02, Clifton, New Jersey
  - Study Site 04, North Charleston, South Carolina
  - Study Site 05, Jackson, Tennessee
  - Study Site 09, Houston, Texas
  - Study Site 10, Katy, Texas
- Bulgaria (7):
  - Study Site 01, Plovdiv
  - Study Site 06, Plovdiv
  - Study Site 02, Sofia
  - Study Site 04, Sofia
  - Study Site 07, Sofia
  - Study Site 05, Stara Zagora
  - Study Site 03, Varna
- Canada (2):
  - Study Site 02, Rimouski, Quebec
  - Study Site 01, Saint-Jérôme, Quebec
- Czechia (9):
  - Study Site 03, Bruntál
  - Study Site 05, Ostrava
  - Study Site 01, Prague
  - Study Site 04, Prague
  - Study Site 08, Prague
  - Study Site 09, Prague
  - Study Site 02, Uherské Hradiště
  - Study Site 07, Uherské Hradiště
  - Study Site 06, Zlín
- Study Site 01, Tallinn, Estonia
- Germany (5):
  - Study Site 03, Berlin
  - Study Site 04, Frankfurt
  - Study Site 06, München
  - Study Site 02, Ratingen
  - Study Site 01, Zerbst
- Hungary (6):
  - Study Site 03, Balatonfüred
  - Study Site 02, Budapest
  - Study Site 04, Budapest
  - Study Site 05, Budapest
  - Study Site 06, Gyula
  - Study Site 01, Veszprém
- Lithuania (2):
  - Study Site 01, Kaunas
  - Study Site 02, Vilnius
- Mexico (5):
  - Study Site 06, León, Guanajuato
  - Study Site 05, Mexico City, Mexico City
  - Study Site 08, Mexico City, Mexico City
  - Study Site 02, Chihuahua City
  - Study Site 03, Distrito Federal
- Poland (10):
  - Study Site 08, Bialystok
  - Study Site 05, Bydgoszcz
  - Study Site 10, Elblag
  - Study Site 04, Gdynia
  - Study Site 02, Katowice
  - Study Site 03, Krakow
  - Study Site 06, Krakow
  - Study Site 09, Poznan
  - Study Site 01, Warsaw
  - Study Site 07, Warsaw
- Russia (11):
  - Study Site 08, Kemerovo
  - Study Site 11, Kemerovo
  - Study Site 04, Kursk
  - Study Site 03, Moscow
  - Study Site 07, Moscow
  - Study Site 10, Moscow
  - Study Site 05, Omsk
  - Study Site 09, Saratov
  - Study Site 06, Smolensk
  - Study Site 01, Tomsk
  - Study Site 02, Yaroslavl
- Serbia (4):
  - Study Site 01, Belgrade
  - Study Site 02, Belgrade
  - Study Site 04, Belgrade
  - Study Site 03, Niška Banja
- Slovakia (5):
  - Study Site 03, Bratislava
  - Study Site 04, Kosice - Saca
  - Study Site 05, Lučenec
  - Study Site 02, Považská Bystrica
  - Study Site 01, Rimavská Sobota
- Ukraine (9):
  - Study Site 08, Donetsk
  - Study Site 01, Kharkiv
  - Study Site 02, Kharkiv
  - Study Site 03, Kyiv
  - Study Site 04, Kyiv
  - Study Site 05, Vinnytsia
  - Study Site 06, Vinnytsia
  - Study Site 07, Vinnytsia
  - Study Site 09, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Vollenhoven RF, Keystone EC, Strand V, Pacheco-Tena C, Vencovsky J, Behrens F, Racewicz A, Zipp D, Rharbaoui F, Wolter R, Knierim L, Schmeidl R, Zhou X, Aigner S, Dalken B, Wartenberg-Demand A; TREAT2b study team. Efficacy and safety of tregalizumab in patients with rheumatoid arthritis and an inadequate response to methotrexate: results of a phase IIb, randomised, placebo-controlled trial. Ann Rheum Dis. 2018 Apr;77(4):495-499. doi: 10.1136/annrheumdis-2017-212478. Epub 2018 Jan 17. PMID 29343509

RESULTS

PARTICIPANT FLOW:
Period: Main Phase I
Arm/Group | Dose Level 1 Tregalizumab | Dose Level 2 Tregalizumab | Dose Level 3 Tregalizumab | Placebo
Started | 83 | 80 | 78 | 80
Completed | 72 | 70 | 70 | 72
Not Completed | 11 | 10 | 8 | 8
Period: Main Phase II
Arm/Group | Dose Level 1 Tregalizumab | Dose Level 2 Tregalizumab | Dose Level 3 Tregalizumab | Placebo
Started | 64 (Non-responders were switched to higher dose Level after Main Phase 1, started = completed -switched.) | 75 (started Patient = completed patients + switched patients (non-responder) from other arms.) | 98 (started Patient = completed patients + switched patients (non-responder) from other arms.) | 44 (non-responders were switched to higher dose Level after Main Phase 1, started = completed -switched)
Completed | 55 | 66 | 76 | 43
Not Completed | 9 | 9 | 22 | 1
Period: Extension Phase
Arm/Group | Dose Level 1 Tregalizumab | Dose Level 2 Tregalizumab | Dose Level 3 Tregalizumab | Placebo
Started | 54 (Some patients terminated or were switched to higher dose Level after Main Phase 2.) | 56 (Some patients terminated or were switched to higher dose Level after Main Phase 2.) | 68 (Some patients terminated after Main Phase 2.) | 0 (No Placebo arm for Extension Phase, all patients terminated or were switched to tregalizumab Groups.)
Completed | 41 | 38 | 44 | 0
Not Completed | 13 | 18 | 24 | 0

BASELINE CHARACTERISTICS:
Population: 8 subjects of 321 who had no post-baseline assessment were excluded from the Full Analysis Set (FAS), (one subject [1.3%] in the placebo group, three subjects [3.6%] in Dose Level 1 Tregalizumab group, two subjects [2.5%] in Dose Level 2 Tregalizumab group, and two subjects [2.6%] in Dose Level 3 Tregalizumab group).
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 Tregalizumab | Dose Level 2 Tregalizumab | Dose Level 3 Tregalizumab | Placebo | Total
Number analyzed (Participants) | 80 | 78 | 76 | 79 | 313
Age, Customized [Number; unit: years]
  0-<40 years | 9 | 19 | 12 | 10 | 50
  40-<=65 years | 62 | 56 | 56 | 57 | 231
  >65 years | 9 | 3 | 8 | 12 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 68 | 58 | 66 | 263
  Male | 9 | 10 | 18 | 13 | 50

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Who Achieve an ACR20 at Week 12 Following Treatment With Tregalizumab + MTX Compared With Subjects Treated on Placebo + MTX
Description: The primary efficacy variable was the proportion of subjects with an ACR20 response after 12 weeks of double-blind treatment with the study medication.
  The analysis of the primary endpoint was performed using observed cases (OC) on the FAS.
Time Frame: Week 12
Population: The analysis of the primary endpoint was performed using observed cases (OC) on the FAS.
  Full analysis set (FAS): All subjects entered into the study who received at least one dose of study medication and have at least one post-baseline assessment.
Measure: Number; unit: percentage of Subjects
Arm/Group | Dose Level 1 Tregalizumab | Dose Level 2 Tregalizumab | Dose Level 3 Tregalizumab | Placebo
Number analyzed (Participants) | 71 | 66 | 70 | 71
percentage of Subjects | 42.3 | 47.0 | 44.3 | 35.2

2. Secondary Outcome: Proportions of Subjects With an ACR 20 Response.
Time Frame: Week 24
Reporting Status: Not Posted

3. Secondary Outcome: Proportions of Subjects With an ACR 50 & 70 Response.
Time Frame: Week 12 & Week 24
Reporting Status: Not Posted

4. Secondary Outcome: Proportions of Subjects With an Disease Activity Score DAS28 <2.6
Time Frame: Week 12 & Week 24
Reporting Status: Not Posted

5. Secondary Outcome: Proportions of Subjects With Low Disease Activity DAS28 ≤3.2
Time Frame: Week 12 & Week 24
Reporting Status: Not Posted

6. Secondary Outcome: ACR Score
Time Frame: up to 48 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Simple Disease Activity Index [SDAI] ≤11
Time Frame: week 12 & 24
Reporting Status: Not Posted

8. Secondary Outcome: Clinical Disease Activity Index [CDAI] ≤10
Time Frame: week 12 & 24
Reporting Status: Not Posted

9. Secondary Outcome: DAS28
Time Frame: up to 48 weeks
Reporting Status: Not Posted

10. Secondary Outcome: EULAR Response
Time Frame: up to 48 weeks
Reporting Status: Not Posted

11. Secondary Outcome: ACR Score Individual Components
Time Frame: up to 48 weeks
Reporting Status: Not Posted

12. Secondary Outcome: DAS28 Score Individual Components
Time Frame: up to 48 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Pharmacokinetics
Description: AUC, Cmax, Tmax at baseline, and at Week (W) 2/Visit (V) 4, W4/V5, W8/V7, W12/V8, W24/V10, W3/V122, W48 (end of Treatment [EoT]/ early termination ET), and at follow-up (post EoT/post ET).
Time Frame: up to 48 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Evaluation of Safety, Patient Reported Outcomes & Blood Tests.
Time Frame: up to 48 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: through study completion, up to 1 year
Description: All adverse events have been matched in accordance with the dosing under which they occurred. This resulted in a higher number of subjects at risk, because some subjects received two dosages. Patients who responded at week 12 continued the same treatment for 12 weeks and non-responders at week 12 were escalated to the next higher dose level or re-randomized to active treatment (placebo patients). After 24 weeks, placebo patients were switched to active treatment during the Extension Phase.
Groups:
- 25mg Dose Level 1 Tregalizumab: Dose Level 1 Tregalizumab (25mg)
- 100mg Dose Level 2 Tregalizumab: Dose Level 2 Tregalizumab (100mg)
- 200mg Dose Level 3 Tregalizumab: Dose Level 3 Tregalizumab (200mg)
- Placebo: Placebo -
Arm/Group | 25mg Dose Level 1 Tregalizumab | 100mg Dose Level 2 Tregalizumab | 200mg Dose Level 3 Tregalizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 3/105 | 1/117 | 7/122 | 1/80
Other Adverse Events (participants affected / at risk) | 14/105 | 16/117 | 15/122 | 9/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25mg Dose Level 1 Tregalizumab (N=105) | 100mg Dose Level 2 Tregalizumab (N=117) | 200mg Dose Level 3 Tregalizumab (N=122) | Placebo (N=80)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple Injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flavivirus Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple Sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Frostbite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lichen Planus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25mg Dose Level 1 Tregalizumab (N=105) | 100mg Dose Level 2 Tregalizumab (N=117) | 200mg Dose Level 3 Tregalizumab (N=122) | Placebo (N=80)
Nasopharyngitis (Infections and infestations) | 7 (9) | 6 (7) | 7 (10) | 4 (4)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6) | 5 (5) | 2 (3)
Headache (Nervous system disorders) | 3 (4) | 6 (9) | 6 (6) | 3 (3)

LIMITATIONS AND CAVEATS:
Due to the lack of efficacy the Extension Phase of the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days